CLINICAL TRIAL: NCT04967547
Title: Effect of Pre-emptive Assessment of Self-care Peritoneal Dialysis (PD) Ability on PD Choice in Patients With Stage 5 Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Na Jiang, Department of Nephrology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: self-care PD ability
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Chronic Kidney Disease (CKD) Stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): be evaluated by using the self-care PD feasibility assessment in addition to education on renal replacement therapy and dialysis
  Interventions: Other: Self-care PD ability assessment form; Other: Education
- Control group (Active Comparator): education on renal replacement therapy and dialysis
  Interventions: Other: Education

INTERVENTIONS:
Other: Self-care PD ability assessment form — Subjects will be evaluated using the self-care PD feasibility assessment tool within 7 days after randomization. The evaluation results will be provided to the patient on the same day
  Arms: Intervention group
Other: Education — Education on renal replacement therapy and dialysis

SUMMARY:
Peritoneal dialysis is an effective renal replacement therapy with higher quality of life and lower treatment cost than hemodialysis.However, the application rate of peritoneal dialysis is much lower than that of hemodialysis. One of the reasons is that patients need to complete fluid changing operation independently, which is especially challenging for elderly and frail patients. Assisted peritoneal dialysis can help patients with independent dialysis disorders to complete dialysis. Currently, there is a lack of standard tools to assess patients' ability to conduct independent dialysis and to determine whether assisted dialysis is needed. Moreover, routine assessment is arranged after the training of dialysis operation, which leads to some patients giving up the procedure at an early stage, resulting in a low selection rate of the procedure.The purpose of this study was to investigate the effect of using a standard scale to evaluate the ability to perform abdominal dialysis in patients with stage 5 chronic kidney disease (CKD) before deciding on dialysis modality.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years old;
2. Need dialysis within 6 months;
3. Informed consent.

Exclusion Criteria:

1. Absolute PD contraindications;
2. Need urgent dialysis;
3. RTX as initial renal replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of PD choice | up to 90 days

SECONDARY OUTCOMES:
The aPD utilization rate | up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fang, MD, Study Director — RenJi Hospital
Locations (1):
- Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China